CLINICAL TRIAL: NCT07304466
Title: Comparison of the Effects of Terlipressin and Somatostatin on Portal Pressure in Patients Undergoing Living Donor Liver Transplantation
Brief Title: Effects of Terlipressin and Somatostatin on Portal Pressure in Patients Undergoing Living Donor Liver Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 6
Record Dates: First submitted 2025-11-24; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplantation; Portal Hypertension
Keywords: liver transplantation; portal pressure; portal hypertension; living donor liver transplantation; somatostatin; terlipressin
MeSH Terms: conditions — Hypertension, Portal | interventions — Somatostatin; Terlipressin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeons performing the portal pressure measurements and the participants will be blinded to group allocation. The study drugs will be prepared and labeled by an independent anesthesiologist/pharmacist not involved in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Somatostatin (SS) (Active Comparator): Somatostatin will be given.
  Interventions: Drug: Somatostatin
- Group Terlipressin (TR) (Active Comparator): Terlipressin will be given.
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Somatostatin — Following baseline portal pressure measurement from the portal vein (25 Gauge intracath, Bıçakçılar®) (PVP0), somatostatin (Somatex®) will be administered as a 250 mcg bolus over 2 minutes, followed by a continuous infusion at 2.5 mcg/kg/hour. Direct portal measurements will be done at the time points explained in the study description.
  Intraoperative ultrasound (GE Healthcare®, linear probe) will be used to record arterial and portal flow parameters. Hemodynamic data will be collected during all measurements. The study drug will be infused continuously for at least 24 hours.
  Arms: Group Somatostatin (SS)
Drug: Terlipressin — Following baseline portal pressure measurement from the portal vein (25 Gauge intracath, Bıçakçılar®) (PVP0), terlipressin (Glypressin®) will be administered as a 1 mg bolus over 2 minutes, followed by a continuous infusion at 2 mcg/kg/hour.
  Direct portal measurements will be done at the time points explained in the study description.
  Intraoperative ultrasound (GE Healthcare®, linear probe) will be used to record arterial and portal flow parameters. Hemodynamic data will be collected during all measurements. The study drug will be infused continuously for at least 24 hours, and up to 5 days if portal pressure remains elevated.
  Arms: Group Terlipressin (TR)

SUMMARY:
The goal of this clinical trial is to compare the effects of somatostatin and terlipressin on lowering portal pressure in patients with portal hypertension undergoing liver transplantation, and to investigate whether there are differences in clinical outcomes between the two drugs. The study will evaluate the decrease in portal pressure from baseline following drug administration at defined time points. It will also compare the effects of these drugs on hemodynamics, bleeding, and transfusion requirements. After baseline intraoperative direct portal pressure measurement, a bolus dose of the study drug will be administered, followed by continuous intravenous infusion intraoperatively and for 24 hours postoperatively. Direct portal pressure will be measured again 5 minutes after the bolus dose, after the portal vein anastomosis, after the hepatic artery anastomosis, and, if performed after splenic artery ligation. Hemodynamic parameters will be recorded, and the drugs will be compared in terms of their intraoperative hemodynamic effects. As elevated portal pressure is associated with increased bleeding, intraoperative blood loss and transfusion needs will also be assessed between the groups. Patients will be followed for 7 days postoperatively for clinical and laboratory outcomes.

DETAILED DESCRIPTION:
It is well known that elevated portal pressure during liver resection is associated with increased bleeding, greater surgical difficulty, impaired splanchnic perfusion, a higher incidence of postoperative kidney injury, and increased need for blood transfusion. Somatostatin, a peptide hormone used to reduce portal pressure, lowers portal venous pressure by altering splanchnic blood flow. It is frequently administered in patients with end-stage liver disease for indications such as controlling variceal bleeding and reducing intraoperative portal pressure. Terlipressin, a vasopressin analog, induces vasoconstriction, thereby decreasing portal inflow and venous congestion in the splanchnic circulation. By lowering portal pressure and exerting favorable systemic effects, it is often used intraoperatively in patients with impaired renal function. It has been associated with reduced surgical bleeding and improved renal perfusion.

Following baseline portal pressure measurement from the portal vein (PVP0), patients will receive treatment according to their study group. In the somatostatin (SS) group, a bolus dose of 250 mcg will be administered over 2 minutes, followed by a maintenance infusion at 2.5 mcg/kg/hour. In the terlipressin (TRP) group, a bolus dose of 1 mg will be given over 2 minutes, followed by a maintenance infusion at 2 mcg/kg/hour. Five minutes after completion of the bolus dose, portal pressure will be measured again and recorded with the corresponding time point (PVP1).

Once the hepatic and portal vein anastomoses are completed and graft reperfusion is achieved, the third portal pressure measurement will be taken (PVP2), and right after completion of the arterial anastomosis, the fourth portal pressure measurement will be performed (PVP3). If PVP exceeds 20 mmHg or Hepatic Venous Pressure Gradient (HVPG) exceeds 15 mmHg, splenic artery ligation will be performed to modify portal inflow and prevent small-for-size syndrome. If performed, this intervention will be recorded, and subsequent measurements will be repeated (PVP4)

Intraoperative ultrasound routinely performed by radiology will be used to measure arterial (peak systolic velocity, resistive index, acceleration time) and portal (flow volume) flow parameters, which will be documented. Hemodynamic data will be recorded throughout all measurements. The study drugs will be administered as continuous infusion for at least 24 hours, and if portal pressure remains elevated, the infusion may be extended up to a maximum of 5 days.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for right lobe living donor liver transplantation with clinically significant portal hypertension (esophageal varices, thrombocytopenia (<100,000), ascites, encephalopathy; Child-Turcotte-Pugh class B-C)

Exclusion Criteria:

* Allergy to any of the medications to be used
* Portal vein thrombosis
* Being treated with terlipressin with a diagnosis of hepatorenal syndrome
* Portopulmonary hypertension
* Acute on chronic liver failure
* Chronic renal failure (glomerular filtration rate ≤ 30%)
* Myocardial ischemia
* Uncontrolled hypertension
* Arrhythmia
* Multiple solid organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Decrease in portal pressure by 20% from the baseline | Baseline (before bolus drug administration) 5 minutes after bolus drug administration Immediately after completion of the portal vein anastomosis Immediately after completion of the hepatic artery anastomosis
  The proportion of patients achieving a ≥20% reduction in portal pressure from baseline at any of the predefined intraoperative assessment timepoints will be recorded.

SECONDARY OUTCOMES:
Change in Portal Pressure (mmHg) | Intraoperative: baseline and subsequent measurements at 5 minutes after bolus administration and immediately after completion of portal and hepatic artery anastomoses.
  The change in portal pressure from baseline will be recorded at predefined intraoperative timepoints using direct portal pressure measurements. The change will be expressed in millimetres of mercury (mmHg).
Amount of bleeding (milliliters) | Periprocedural
  Total intraoperative blood loss will be measured in millilitres.
Perioperative Blood Transfusion (Units) | During the perioperative period
  The total number of blood units transfused during the perioperative period will be recorded.
Hepatic Artery Peak Systolic Flow (cm/s) | Immediately after arterial anastomosis (intraoperative)
  The peak systolic flow of the hepatic artery will be measured by intraoperative Doppler ultrasound after completion of the arterial anastomosis.
Portal Vein Flow Velocity (cm/s) | Immediately after completion of the hepatic arterial anastomosis (intraoperative)
  Portal vein flow velocity will be measured intraoperatively using Doppler ultrasound immediately after completion of the hepatic arterial anastomosis. The value will be recorded as a single measurement in centimetres per second (cm/s).
Hepatic artery acceleration time (AT). | Immediately after completion of the hepatic arterial anastomosis (intraoperative
  Hepatic artery acceleration time (milliseconds) will be measured using Doppler ultrasound immediately after completion of the hepatic artery anastomosis to evaluate arterial waveform characteristics and early graft inflow dynamics.
Splenic Artery Ligation (Yes/No) | During the intraoperative period
  Whether splenic artery ligation is performed during the transplant surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ayşe ince, Principal Investigator — Istanbul Medipol University Medipol Mega Hospital

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data (IPD).

REFERENCES:
- [Background] Mahdy MM, Abbas MS, Kamel EZ, Mostafa MF, Herdan R, Hassan SA, Hassan R, Taha AM, Ibraheem TM, Fadel BA, Geddawy M, Sayed JA, Ibraheim OA. Effects of terlipressin infusion during hepatobiliary surgery on systemic and splanchnic haemodynamics, renal function and blood loss: a double-blind, randomized clinical trial. BMC Anesthesiol. 2019 Jun 15;19(1):106. doi: 10.1186/s12871-019-0779-6. PMID 31200638
- [Background] Li XL, Zhu XD, Xiao N, Liu XF, Xu B, Shi GM, Huang C, Shen YH, Cai JB, Zhou J, Fan J, Sun HC. A prospective study of the effect of terlipressin on portal vein pressure and clinical outcomes after hepatectomy: A pilot study. Surgery. 2020 Jun;167(6):926-932. doi: 10.1016/j.surg.2020.01.013. Epub 2020 Feb 26. PMID 32113581
- [Background] Papaluca T, Gow P. Terlipressin: Current and emerging indications in chronic liver disease. J Gastroenterol Hepatol. 2018 Mar;33(3):591-598. doi: 10.1111/jgh.14009. PMID 28981166
- [Background] Abraldes JG, Bosch J. Somatostatin and analogues in portal hypertension. Hepatology. 2002 Jun;35(6):1305-12. doi: 10.1053/jhep.2002.33469. No abstract available. PMID 12029614
- [Background] Lizaola-Mayo B, Vargas HE. Hepatorenal Syndrome-Acute Kidney Injury in Liver Transplantation. Clin Gastroenterol Hepatol. 2023 Sep;21(10S):S20-S26. doi: 10.1016/j.cgh.2023.06.010. PMID 37625863
- [Background] Iwakiri Y. Pathophysiology of portal hypertension. Clin Liver Dis. 2014 May;18(2):281-91. doi: 10.1016/j.cld.2013.12.001. Epub 2014 Feb 25. PMID 24679494
- [Background] Giabicani M, Joly P, Sigaut S, Timsit C, Devauchelle P, Dondero F, Durand F, Froissant PA, Lamamri M, Payance A, Restoux A, Roux O, Thibault-Sogorb T, Valainathan SR, Lesurtel M, Rautou PE, Weiss E. Predictive role of hepatic venous pressure gradient in bleeding events among patients with cirrhosis undergoing orthotopic liver transplantation. JHEP Rep. 2024 Feb 28;6(6):101051. doi: 10.1016/j.jhepr.2024.101051. eCollection 2024 Jun. PMID 38699073